CLINICAL TRIAL: NCT04156269
Title: Phase I, Interventional, Single Arm, Open Label, Treatment Study to Evaluate the Safety and Tolerability of BCMA-CS1 cCAR in Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: BCMA-CS1 Compound CAR (cCAR) T Cells for Relapsed/Refractory Multiple Myeloma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: iCell Gene Therapeutics (Industry)
Collaborators: Peking University Shenzhen Hospital (Other); Chengdu Military General Hospital (Other); iCAR Bio Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICG182-001
Record Dates: First submitted 2019-11-06; First posted 2019-11-07 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-01

CONDITIONS: Multiple Myeloma
Keywords: BCMA; CS1; BCMA-CS1 cCAR T cells; CD269; SLAMF7
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCMA-CD33 cCAR T cells (Experimental): BCMA-CS1 cCAR T cells transduced with a lentiviral vector to express two distinct units of anti-BCMA and CS1 CARs
  Interventions: Biological: BCMA-CS1 cCAR T cells

INTERVENTIONS:
Biological: BCMA-CS1 cCAR T cells — BCMA-CS1 cCAR T cells administered to patients, will be either fresh or thawed CAR T cells by IV injection after receiving lymphodepleting chemotherapy.

SUMMARY:
This is a phase I, interventional, single arm, open label, treatment study to evaluate the safety and tolerability of BCMA-CS1 cCAR in patients with relapsed and/or refractory multiple myeloma.

DETAILED DESCRIPTION:
BCMA-CS1 cCAR (Compound CAR BCMA-CS1) is a chimeric antigen receptor immunotherapy treatment designed to treat multiple myeloma using two different antigen targets, BCMA (CD269) and CS1 (SLAMF7).

The use of two different targets widely expressed on plasma cells, BCMA and CS1, intends to increase coverage and eradicate cancerous cells before resistance develops in surviving cancer cells that have undergone selective pressures or antigen escape. BCMA-CS1 cCAR bears two distinct functional CAR molecules expressed on a T-cell, directed against the surface proteins BCMA and CS1.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis based on the World Health Organization (WHO) 2008
2. Patients have exhausted standard therapeutic options
3. Systematic usage of immunosuppressive drug or corticosteroid must have been stopped for more than 4 weeks
4. Female must be not pregnant during the study

Exclusion Criteria:

1. Prior solid organ transplantation
2. Potentially curative therapy including chemotherapy or hematopoietic cell transplant
3. Prior treatment with BCMAxCD3 or CS1xCD3 bispecific agents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-08-31 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicity (DLT) as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | 28 days
Type of dose-limiting toxicity (DLT) | 28 days
Number of participants with adverse event by severity as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | 2 years

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 1 year
  Assessment of morphologic complete remission (CR), complete remission with incomplete recovery of counts (CR1), no residual disease as analyzed by flow cytometry analysis, and molecular remission by molecular studies
Progression-free survival (PFS) | 1 year
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hongyu Zhang, MD, PhD, Principal Investigator — Peking University Shenzhen Hospital; Fang Liu, MD, PhD, Principal Investigator — Chengdu Military General Hospital
Locations (2):
- China (2):
  - Chengdu Military General Hospital, Chengdu
  - Peking University Shenzhen Hospital, Shenzhen

IPD SHARING:
Plan to Share IPD: No